CLINICAL TRIAL: NCT06710327
Title: Effect of Tranexamic Acid on Intraoperative Blood Loss in Patients Undergoing Aquablation for Benign Prostatic Hyperplasia: a Randomized Controlled Trial
Brief Title: Effect of Tranexamic Acid on Intraoperative Blood Loss in Patients Undergoing Aquablation
Acronym: TXA-AQ
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: KPSC IRB 056236; KPSC IRB 056263 (Other: Kaiser Permanente Southern California IRB)
Record Dates: First submitted 2024-11-22; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: BPH; TXA; Aquablation; Benign Prostatic Hyperplasia; Tranexamic Acid
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive an intravenous (IV) administration of a placebo prior to their Aquablation procedure. This placebo is a saline solution that looks identical to the tranexamic acid (TXA) used in the Intervention Group but contains no active medication. The placebo is given to mimic the administration of TXA to ensure that the study conditions are the same for both groups, except for the active treatment. All other aspects of the surgical procedure and postoperative care remaining standardized across both study arms.
  Interventions: Drug: Placebo
- TXA Administration (Experimental): Participants receive tranexamic acid (TXA) preoperatively via intravenous (IV) administration. The dose consists of 1g of TXA delivered in a single IV push immediately prior to the Aquablation therapy. TXA acts as an antifibrinolytic agent, preventing excessive blood loss by stabilizing the formation of blood clots during surgery. This intervention aims to assess TXA's efficacy in reducing perioperative blood loss compared to placebo, with all other aspects of the surgical procedure and postoperative care remaining standardized across both study arms.
  Interventions: Drug: Tranexamic Acid (IV)

INTERVENTIONS:
Drug: Tranexamic Acid (IV) — The intervention is administered as a clear, colorless solution infusion. The dosage administered is a 1 gram intravenous (IV) push, delivered immediately before starting the Aquablation therapy. The administration of TXA occurs only once, as a single dose preoperatively.
  Other Names: TXA; Cyclokapron
  Arms: TXA Administration
Drug: Placebo — Participants receive a saline solution, which is a sodium chloride (0.9%) IV infusion, identical in appearance to the TXA solution. The saline is administered as a single 1 gram-equivalent volume intravenous (IV) push, delivered immediately before the Aquablation therapy commences. This singular administration matches the frequency and timing of the TXA intervention to ensure uniformity across both study groups, maintaining the blinding of the study.
  Other Names: normal saline; NS
  Arms: Placebo

SUMMARY:
This study aims to find out if tranexamic acid (TXA), a medication, works to decrease blood loss during a specific surgery called Aquablation therapy, which is a treatment for men with Benign Prostatic Hyperplasia (BPH). BPH is a common condition in men over the age of 45 that involves enlargement of the prostate gland and can lead to problems or discomfort with urination.

The main goal of this research is to see if TXA can help reduce the amount of blood loss during surgery compared to not using the drug. This is important because losing less blood during surgery can help patients recover faster and more safely. Researchers will monitor the safety of TXA and its effects on other outcomes, like the length of hospital stay and any possible changes in blood tests that check how well blood clots.

Participants in this study will:

* Be males diagnosed with BPH who are already scheduled to undergo Aquablation therapy.
* Be randomly assigned to either receive TXA or a placebo (a look-alike substance that contains no drug) right before their surgery.
* Not know which treatment they are receiving to make sure the results are unbiased.

Researchers hope to engage participants who meet the health criteria of the study. They will be carefully monitored before, during, and after the surgery for any health changes, and their blood loss during surgery will be measured.

This study does not require any additional time commitment outside of the standard surgical process, and all treatments will be provided at no additional cost to the participants. The researchers will ensure that all participants understand the procedure and support their safety throughout the research.

DETAILED DESCRIPTION:
This clinical study is investigating whether a medication called tranexamic acid (TXA) can help reduce blood loss during a type of prostate surgery known as Aquablation therapy. This therapy is used to treat Benign Prostatic Hyperplasia (BPH), a common condition in older men that results in the enlargement of the prostate gland which can cause difficulty with urination.

Purpose of the Study:

The primary purpose of this research is to determine if TXA makes this surgery safer by decreasing the amount of blood lost during the procedure. Reducing blood loss during surgery is beneficial because it can lead to quicker recovery times and reduce the likelihood of complications. The study will also look at other important factors such as the overall safety of using TXA, its effect on the length of time participants stay in the hospital after surgery, and whether it causes any significant changes in blood clotting tests.

How the Research Will Happen:

Participants in the study will be men diagnosed with BPH who are planning to undergo Aquablation therapy. They will be randomly placed into one of two groups:

One group will receive TXA through an IV right before their surgery. The other group will receive a placebo, which is a substance that looks like the medication but contains no active drug, administered in the same way.

This setup ensures that neither the participants nor the health care providers know who receives the TXA and who receives the placebo, helping to maintain objectivity in the results.

What Participants Will Do:

Participants will visit the hospital as they normally would for their scheduled surgery. Before the surgery, they will receive either TXA or the placebo. The procedure itself and the immediate recovery process do not change. Researchers will collect information about how much blood participants lose during surgery and monitor their recovery closely.

The number of visits and what each participant needs to do during the study remains the same as what would happen during typical Aquablation therapy. Besides receiving the TXA or placebo, there are no additional procedures or drugs involved.

Safety Measures:

Study researchers are committed to participant safety. Participants will be closely monitored throughout the surgery and their recovery. The research team will watch for any side effects or reactions to the medication, especially any signs of blood clotting or allergic reactions, as TXA is known to affect blood clotting. If there are any concerns about a participant's health, they can be quickly addressed by the medical team.

Why This Matters:

For men undergoing Aquablation therapy for BPH, managing blood loss is a major safety concern. If TXA can effectively reduce blood loss without causing other complications, it could improve the outcomes for thousands of men who undergo this surgery every year.

This study will help doctors better understand the benefits and risks of using TXA in this setting, potentially leading to its wider use in similar surgeries to improve patient safety and outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants diagnosed with BPH scheduled for Aquablation therapy.
2. Aged 45 years or older
3. Exhibiting clinically significant symptoms of BPH.

Exclusion Criteria:

1. History of or high risk for thrombosis.
2. Presence of preoperative heart or cerebrovascular diseases.
3. Renal insufficiency.
4. Ongoing anticoagulation therapy.
5. Required extended preoperative resting period.
6. Diagnosis of prostate cancer.
7. Any form of blood coagulation dysfunction.
8. Previous use of warfarin or aspirin before the surgery.
9. Belonging to vulnerable populations such as prisoners (who are not treated in our clinics).

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Perioperative Hemoglobin Change | Measured preoperatively and postoperatively, within 2 hours of surgery completion
  The primary outcome measure is the efficacy of tranexamic acid (TXA) in decreasing the amount of hemoglobin lost during Aquablation therapy compared to placebo. This will be quantitatively assessed by measuring the hemoglobin levels in patients' blood samples collected immediately before and after the procedure. The change in hemoglobin levels will be compared between the TXA-treated group and the placebo group to determine if TXA administration results in a significantly smaller decrease in hemoglobin, indicating less blood loss.

SECONDARY OUTCOMES:
Rate of Perioperative Complications Associated with Tranexamic Acid | From initiation of surgery to post-operative follow up, up to 60 days post-surgery.
  This measure tracks the incidence of perioperative complications, including but not limited to thromboembolic events, which are potential risks associated with TXA. The frequency of these complications will be compared between patients treated with TXA and those receiving a placebo to understand any increased risks when using TXA in the context of Aquablation therapy.
Length of Hospital Stay Post-Aquablation Therapy | From time of surgery to hospital discharge, typically within 1 day post-surgery
  This secondary outcome evaluates whether TXA administration affects the length of postoperative hospital stay compared to placebo. The length of stay is calculated from the time of surgery completion to the time of discharge, aiming to ascertain if TXA can contribute to a faster recovery and shorter hospitalization.
Change in ProThrombin Time (PT) Following Tranexamic Acid Administration | Lab values measured preoperatively and within 2 hours post-surgery.
  This measure determines if TXA administration has any significant effect on an element of the coagulation, prothrombin time (PT). Serum sample will be collected and analyzed preoperatively and postoperatively to detect any changes that might indicate a heightened risk of clotting or bleeding abnormalities.
Change in activated partial thromboplastin time (aPTT) Following Tranexamic Acid Administration | Lab values measured preoperatively and within 2 hours post-surgery.
  This measure determines if TXA administration has any significant effect on an element of the coagulation, activated partial thromboplastin time (aPTT). Serum sample will be collected and analyzed preoperatively and postoperatively to detect any changes that might indicate a heightened risk of clotting or bleeding abnormalities.
Change in activated fibrinogen level Following Tranexamic Acid Administration | Lab values measured preoperatively and within 2 hours post-surgery.
  This measure determines if TXA administration has any significant effect on an element of the coagulation and platelet activity, fibrinogen. Serum sample will be collected and analyzed preoperatively and postoperatively to detect any changes that might indicate a heightened risk of clotting or bleeding abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher F Tenggardjaja, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Los Angeles Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data from this study will not be shared publicly due to concerns regarding participant privacy and confidentiality. The sensitivity of the health information collected, especially in a clinical trial context, requires strict adherence to privacy protections. Disclosure risks associated with sharing detailed IPD can potentially lead to identification of participants, despite data anonymization procedures.
  Furthermore, the consent forms participants will sign at the beginning of the trial include clauses that specifically limit the use of their data to the researchers involved in this study and for the purpose of assessing the efficacy and safety of tranexamic acid in this specific surgical setting. As such, participants will not be consented to broader data sharing with the public or external entities.